CLINICAL TRIAL: NCT06074458
Title: GO TEAM INTERVENTION PROTOCOL: GLUCOSE OPTIMIZATION THROUGH TECHNOLOGY ASSISTED MANAGEMENT: Use of a Diabetes Dashboard and Community Health Worker to Decrease Disparities in Technology Use in Pediatric T1D
Brief Title: GO TEAM: Glucose Optimization Through Technology Assisted Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah MacLeish (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); KeborMed (Unknown)
Responsible Party: Sponsor-Investigator, Sarah MacLeish, Associate Professor of Pediatrics, Case Western Reserve University
Organization: Case Western Reserve University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Study20230860; 1R01DK134953 (NIH)
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes
Keywords: Pediatric; Diabetes Technology; Disparities
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Participants in this arm follow standard of care procedures.
- Diabetes Dashboard and Community Health Worker (Active Comparator): Participants diabetes technology devices will be linked to a remote patient monitoring dashboard and will have access to a Smartphone application, as well as scheduled and as needed visits with a community health worker.
  Interventions: Other: Glucosano; Behavioral: Community Health Worker diabetes technology coach

INTERVENTIONS:
Other: Glucosano — Glucosano is a remote patient monitoring diabetes dashboard with a patient facing Smartphone application
  Arms: Diabetes Dashboard and Community Health Worker
Behavioral: Community Health Worker diabetes technology coach — Community Health Workers will work with participants as a diabetes technology coach during scheduled and as needed visits
  Arms: Diabetes Dashboard and Community Health Worker

SUMMARY:
Black/African American children and young adults with type 1 diabetes are less likely to use diabetes technologies, such as continuous glucose monitors, insulin pumps, and automated insulin delivery systems, compared to White children and young adults. The investigators are working to find ways to make sure that all patients with type 1 diabetes are equally able to use these technologies. The purpose of this study is to find out if a new computer program for the diabetes team, along with a smartphone app (called Glucosano) for patients/parents, as well as a community health worker, are accepted and used by Black/African American patients and parents living with type 1 diabetes, and if this can help decrease racial disparities in the use of diabetes technologies.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported as Non-Hispanic Black
* Clinical diagnosis of T1D requiring treatment with insulin at the time of consent
* Not currently (within the past 3 months) using an automated insulin delivery system \
* Willingness to wear a continuous glucose monitor for 10 days at 3 different time points, and willingness to consider use of a personal continuous glucose monitor

Exclusion Criteria:

* Clinical diagnosis of Type 2 or monogenic diabetes
* Completed high school
* Non-English speaking guardians
* Automated insulin delivery system use within the past 3 months
* Custody of children and family services

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of participants who start on automated insulin delivery (AID) as measured by medical records review | Baseline, 4 weeks, 3 months, 6 months, 9 months, 12 months
Change in percentage of participants who remain on AID as measured by medical record review | Baseline, 4 weeks, 3 months, 6 months, 9 months, 12 months

SECONDARY OUTCOMES:
Change in patient endorsement of intervention as measured by the Acceptability of Intervention Measure (AIM) | 3 months and 12 months
  4 item measure of acceptability using 5 point Likert scale, where 1 is completely disagree and 5 is completely agree
Change in patient endorsement of intervention as measured by Feasibility of Intervention Measure (FIM) | 3 months and 12 months
  4 item measure of feasibility using 5 point Likert scale, where 1 is completely disagree and 5 is completely agree
Change in patient endorsement of intervention as measured by Intervention Appropriateness Measure (IAM) | 3 months and 12 months
  4 item measure of appropriateness using 5 point Likert scale, where 1 is completely disagree and 5 is completely agree
Number of times patient reached out to team as measured by medical record review | Up to 12 months
Number of automatically generated alerts as measured by dashboard/app review | Up to 12 months
Number of times a physician or diabetes nurse interacted with patient as measured by dashboard review | Up to 12 months
Number of alerts as measured by dashboard review | Up to 12 months
Number of phone calls initiated by patients as measured by dashboard review | Up to 12 months
Number of downloads of the app | Up to 12 months
Number of days of patient/family use interaction with the app as measured by dashboard review | Up to 12 months
Change in percentage of participants using continuous glucose monitor (CGM) with at least 80% wear time as measured by CGM data | Baseline, 4 weeks, 3 months, 6 months, 9 months, 12 months
Change in percentage of CGM wear time as measured by CGM data | Baseline, 4 weeks, 3 months, 6 months, 9 months, 12 months
Change in percentage of participants using an insulin pump as measured by chart review | Baseline, 4 weeks, 3 months, 6 months, 9 months, 12 months
Change in capillary HbA1c | Baseline, 3 months, 6 months, 9 months, 12 months
Change in time in range as measured by continuous glucose monitoring | 4 weeks, 6 months, 12 months
  Time in range is time glucose is between 70-180 mg/dL
Change in time glucose is <70 mg/dL as measured by continuous glucose monitoring | 4 weeks, 6 months, 12 months
Change in time glucose >250 mg/dL as measured by continuous glucose monitoring | 4 weeks, 6 months, 12 months
Psychosocial functioning of children/adolescents, as measured by the strengths and difficulties questionnaire given to parents | Baseline
  25-item questionnaire using a 3-point Likert scale, with one being not true and 3 being certainly true
Change in diabetes family conflict, as measured by the Diabetes Family Conflict Scale | 4 weeks, 12 months
  19-item questionnaire using 3-point Likert scale, where 1 is almost never and 3 is almost always
Change in child/adolescent quality of life, as measured by PedsQL Type 1 diabetes module by parent-proxy | 4 weeks, 12 months
  28-item questionnaire using 5-point Likert scale, where 0 is almost never a problem and 4 is almost always a problem
Change in parental burden related to diabetes, as measured by Problem Areas in Pediatric Diabetes - Parent Revised Version | 4 weeks, 12 months
  18-item questionnaire using 5-point Likert scale, where 0 is agree and 4 is disagree
Change in medical distrust, as measured by the Group Based Medical Distrust Scale | Baseline, 12 months
  12-item questionnaire using 5 point Likert scale, where 1 is strongly disagree and 5 is strongly agree
Change personal frequency of discrimination in healthcare, as measured by the Racism in Healthcare Index | Baseline, 12 months
  7-item questionnaire regarding frequency of discrimination in healthcare ranging from never to 4 times or more in a lifetime
Change in perceptions of racism in healthcare, as measured by the Racism in Healthcare Index | Baseline, 12 months
  4-item questionnaire using 5 point Likert scale where 1 is strongly disagree and 5 is strongly agree
Change in diabetes specific attitudes towards technology as measured by the Diabetes Specific Technology Attitudes Scale | Baseline, 12 months
  5-item questionnaire using 5 point Likert scale, where 1 is strongly disagree and 5 is strongly agree
Change in barriers to technology as measured by Barriers to Technology Checklist | Baseline, 12 months
  19-item yes/no questionnaire
CGM satisfaction as measured by the CGM satisfaction scale | 12 months
  37-item questionnaire using 5-point Likert scale, where 1 is strongly disagree and 5 is strongly agree
Change in diabetes management self-efficacy as measured by the Self-Efficacy for Diabetes Self-Management scale short version | 4 weeks, 12 months
  10-item questionnaire using 6-point Likert scale, where 1 is "very sure I can't" and 6 is "very sure I can"
Benefits and Burdens of CGM as measured by Benefits and Burdens of CGM scale | 12 months
  16-item questionnaire using 5-point Likert scale, where 1 is strongly disagree and 5 is strongly agree
Episodes of Diabetic Ketoacidosis as measured by chart review | up to 12 months
  DKA defined as presence of all of the following: 1) blood glucose greater than 250 mg/dL, 2) pH less than 7.3 OR bicarbonate less 15 mEq/L, 3)Moderate or large ketones in urine OR blood ketone >3 mmol/L, 4) Requiring treatment within a health care facility.
Episodes of severe hypoglycemia as measured by chart review | up to 12 months
  Unconscious or having a seizure due to hypoglycemia

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No